CLINICAL TRIAL: NCT06986876
Title: Exploration of the Perceptions of Women With a History of Gestational Diabetes From the Gonesse Hospital Catchment Area Regarding Their Risk of Developing Type 2 Diabetes.
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Gonesse (Other)
Responsible Party: Sponsor
Other Study IDs: 0093_ENDOCRINOLOGIE
Record Dates: First submitted 2025-05-15; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus, Type 2; Diabetes, Gestational
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study focuses on the patients' perspective and aims to provide explanatory elements regarding the barriers to type 2 diabetes screening among women with a history of gestational diabetes. The main objective is to understand the obstacles and enablers in order to optimize type 2 diabetes screening in women with a history of gestational diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Women with a history of gestational diabetes
* Aged between 18 and 45 years
* French-speaking
* Followed up at Gonesse Hospital

Exclusion Criteria:

* Under 18 or over 45 years old
* Non-French-speaking

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: The study population will consist of women aged 18 to 45 years who have a history of gestational diabetes, are French-speaking, and reside within the catchment area of Gonesse Hospital (Île-de-France region, France). These participants represent a population at increased risk of developing type 2 diabetes and are targeted for better understanding of the barriers and facilitators to post-partum diabetes screening.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Identification and qualitative analysis of the factors influencing participation in type 2 diabetes screening among women with a history of gestational diabetes. | 15 january 2025 - 15 may 2025

CONTACTS AND LOCATIONS:
Locations (1):
- France, Gonesse, France, France